CLINICAL TRIAL: NCT02421926
Title: Extension Study of a Study to Evaluate Efficacy and Safety of Imatinib (Glinib®) 600mg/Day Depending on Early Molecular Response in Newly Diagnosed Patients With Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Extension Study of IDEAL (Imatinib) for Chronic Myelgenous Leukemia (CML)
Acronym: IDEAL-E
Status: Withdrawn | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor, Asan Medical Center
Other Study IDs: H-99
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Dasatinib; 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IDEAL-E observational group: Subjects who were newly diagnosed as chronic phase chronic myelogenous leukemia, were enrolled to 'IDEAL' study, finished the total study period of 'IDEAL' study or were dropped during the study period.
  Interventions: Drug: IDEAL-E observation (investigators choice of imatinib, nilotinib, dasatinib, radotinib)

INTERVENTIONS:
Drug: IDEAL-E observation (investigators choice of imatinib, nilotinib, dasatinib, radotinib) — After the end of follow-up period of IDEAL study, subjects who agree with this extension study (IDEAL-E) will be enrolled and be followed up for additional 4 years to evaluate the duration of treatment response, disease progression, and survival status. Subjects who will be enrolled in this prospective observational study will be treated with drugs - imatinib 300-600mg / nilotinib 600mg / dasatinib 100mg / radotinib 800mg - which has been chosen by the each investigator according to the drug compliance and overall response. The drug choice will be at the discretion of each investigator, and the overall adverse event / molecular response will be monitored every 6 months in this prospective observational study.
  Other Names: glinib, sprycel, tasigna, supect

SUMMARY:
This study is an extension study (prospective observational study) of 'IDEAL' study (A Study to Evaluate Efficacy and Safety of Imatinib (Glinib) 600mg/day depending on Early Molecular Response in Newly Diagnosed Patients with Chronic Myeloid Leukemia in Chronic Phase, NCT02204722) to evaluate the duration of treatment response, disease progression, and survival status up to 5 years after the inclusion.

DETAILED DESCRIPTION:
We have started a prospective study of evaluating efficacy and safety of imatinib 600mg/day depending on early molecular response in newly diagnosed patients with chronic myelogenous leukemia in chronic phase (IDEAL, NCT02204722), which will enroll 150 patients and follow up them for 1 years for the purpose of evaluating the primary endpoints - difference of major molecular response rate at 1 year. However, Chronic myelogenous is a disease which needs long-term for the outcome of treatment with BCR-ABL tyrosine kinase inhibitor. After the end of follow-up period of IDEAL study, subjects who agree with this extension study (IDEAL-E) will be enrolled and be followed up for additional 4 years to evaluate the duration of treatment response, disease progression, and survival status. Subjects who will be enrolled in this prospective observational study will be treated with drugs - imatinib 300-600mg / nilotinib 600mg / dasatinib 100mg - which has been chosen by the each investigator according to the drug compliance and overall response. The drug choice will be at the discretion of each investigator, and the overall adverse event / molecular response will be monitored every 6 months in this prospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were newly diagnosed as chronic phase chronic myelogenous leukemia, were enrolled to 'IDEAL study (A Phase IV Study to Evaluate Efficacy and Safety of Imatinib(Glinib®) 600mg/day Depending on Early Molecular Response in Newly Diagnosed Patients with Chronic Myeloid Leukemia in Chronic Phase, NCT02204722)
* Subjects who agreed with the participation of this study after informed consent

Exclusion Criteria:

* Patients who were newly diagnosed as chronic phase chronic myelogenous leukemia, agree with the participation to 'IDEAL study (A Phase IV Study to Evaluate Efficacy and Safety of Imatinib(Glinib®) 600mg/day Depending on Early Molecular Response in Newly Diagnosed Patients with Chronic Myeloid Leukemia in Chronic Phase, NCT02204722) after informed consent, but were excluded finally from the 'IDEAL' study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were newly dianosed as chronic phase chronic myelogenous leukemia, were enrolled to 'IDEAL' study, and were followed up
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate | 5-year

SECONDARY OUTCOMES:
failure-free survival rate | 2-year
failure-free survival rate | 5-year
cumulative incidence of progression to accelerated phase / blast crisis | 2-year
cumulative incidence of progression to accelerated phase / blast crisis | 5-year
overall survival | 2-year
overall survival | 5-year
progression-free survival rate | 2-year

OTHER OUTCOMES:
cumulative incidence of hematologic adverse events | 2-year
cumulative incidence of hematologic adverse events | 5-year
cumulative incidence of non-hematologic adverse events | 2-year
cumulative incidence of non-hematologic adverse events | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-Hyung Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (12):
- South Korea (12):
  - Seoul National University Bundang Hospital, Seongnam, Gyong-gi Province
  - Korea University Ansan Hospital, Ansan
  - Busan National University Hospital, Busan
  - Haeundae Paik Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchyunhyang University Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Background] Kantarjian HM, Larson RA, Guilhot F, O'Brien SG, Mone M, Rudoltz M, Krahnke T, Cortes J, Druker BJ; International Randomized Study of Interferon and STI571 (IRIS) Investigators. Efficacy of imatinib dose escalation in patients with chronic myeloid leukemia in chronic phase. Cancer. 2009 Feb 1;115(3):551-60. doi: 10.1002/cncr.24066. PMID 19117345
- [Background] Hehlmann R, Lauseker M, Jung-Munkwitz S, Leitner A, Muller MC, Pletsch N, Proetel U, Haferlach C, Schlegelberger B, Balleisen L, Hanel M, Pfirrmann M, Krause SW, Nerl C, Pralle H, Gratwohl A, Hossfeld DK, Hasford J, Hochhaus A, Saussele S. Tolerability-adapted imatinib 800 mg/d versus 400 mg/d versus 400 mg/d plus interferon-alpha in newly diagnosed chronic myeloid leukemia. J Clin Oncol. 2011 Apr 20;29(12):1634-42. doi: 10.1200/JCO.2010.32.0598. Epub 2011 Mar 21. PMID 21422420
- [Background] Hughes TP, Branford S, White DL, Reynolds J, Koelmeyer R, Seymour JF, Taylor K, Arthur C, Schwarer A, Morton J, Cooney J, Leahy MF, Rowlings P, Catalano J, Hertzberg M, Filshie R, Mills AK, Fay K, Durrant S, Januszewicz H, Joske D, Underhill C, Dunkley S, Lynch K, Grigg A; Australasian Leukaemia and Lymphoma Group. Impact of early dose intensity on cytogenetic and molecular responses in chronic- phase CML patients receiving 600 mg/day of imatinib as initial therapy. Blood. 2008 Nov 15;112(10):3965-73. doi: 10.1182/blood-2008-06-161737. Epub 2008 Sep 3. PMID 18768781
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Druker BJ, Guilhot F, O'Brien SG, Gathmann I, Kantarjian H, Gattermann N, Deininger MW, Silver RT, Goldman JM, Stone RM, Cervantes F, Hochhaus A, Powell BL, Gabrilove JL, Rousselot P, Reiffers J, Cornelissen JJ, Hughes T, Agis H, Fischer T, Verhoef G, Shepherd J, Saglio G, Gratwohl A, Nielsen JL, Radich JP, Simonsson B, Taylor K, Baccarani M, So C, Letvak L, Larson RA; IRIS Investigators. Five-year follow-up of patients receiving imatinib for chronic myeloid leukemia. N Engl J Med. 2006 Dec 7;355(23):2408-17. doi: 10.1056/NEJMoa062867. PMID 17151364
- [Background] Baccarani M, Rosti G, Castagnetti F, Haznedaroglu I, Porkka K, Abruzzese E, Alimena G, Ehrencrona H, Hjorth-Hansen H, Kairisto V, Levato L, Martinelli G, Nagler A, Lanng Nielsen J, Ozbek U, Palandri F, Palmieri F, Pane F, Rege-Cambrin G, Russo D, Specchia G, Testoni N, Weiss-Bjerrum O, Saglio G, Simonsson B. Comparison of imatinib 400 mg and 800 mg daily in the front-line treatment of high-risk, Philadelphia-positive chronic myeloid leukemia: a European LeukemiaNet Study. Blood. 2009 May 7;113(19):4497-504. doi: 10.1182/blood-2008-12-191254. Epub 2009 Mar 4. PMID 19264678
- [Background] Piazza RG, Magistroni V, Franceschino A, Andreoni F, Tornaghi L, Colnaghi F, Corneo G, Pogliani EM, Gambacorti-Passerini C. The achievement of durable complete cytogenetic remission in late chronic and accelerated phase patients with CML treated with Imatinib mesylate predicts for prolonged response at 6 years. Blood Cells Mol Dis. 2006 Sep-Oct;37(2):111-5. doi: 10.1016/j.bcmd.2006.06.002. Epub 2006 Aug 14. PMID 16908206
- [Background] Breccia M, Alimena G. The significance of early, major and stable molecular responses in chronic myeloid leukemia in the imatinib era. Crit Rev Oncol Hematol. 2011 Aug;79(2):135-43. doi: 10.1016/j.critrevonc.2010.07.003. Epub 2010 Aug 4. PMID 20685131
- [Background] Baccarani M, Cortes J, Pane F, Niederwieser D, Saglio G, Apperley J, Cervantes F, Deininger M, Gratwohl A, Guilhot F, Hochhaus A, Horowitz M, Hughes T, Kantarjian H, Larson R, Radich J, Simonsson B, Silver RT, Goldman J, Hehlmann R; European LeukemiaNet. Chronic myeloid leukemia: an update of concepts and management recommendations of European LeukemiaNet. J Clin Oncol. 2009 Dec 10;27(35):6041-51. doi: 10.1200/JCO.2009.25.0779. Epub 2009 Nov 2. PMID 19884523
- [Background] Marin D, Ibrahim AR, Lucas C, Gerrard G, Wang L, Szydlo RM, Clark RE, Apperley JF, Milojkovic D, Bua M, Pavlu J, Paliompeis C, Reid A, Rezvani K, Goldman JM, Foroni L. Assessment of BCR-ABL1 transcript levels at 3 months is the only requirement for predicting outcome for patients with chronic myeloid leukemia treated with tyrosine kinase inhibitors. J Clin Oncol. 2012 Jan 20;30(3):232-8. doi: 10.1200/JCO.2011.38.6565. Epub 2011 Nov 7. PMID 22067393